CLINICAL TRIAL: NCT04246112
Title: A Handwriting Intervention Program for Children With Tic Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jan Rowe, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300003428; Departmental funding (Other: UAB, peds neurology)
Record Dates: First submitted 2019-10-14; First posted 2020-01-29 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Tourette Syndrome; Tic Disorders
Keywords: Handwriting; Pediatrics
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Intervention Model Description: A handwriting skills training software program MovAlyzeR® will be given and downloaded to the children's laptop computer. Participants will be requested to use the software program to practice handwriting 15-20 minutes per day, 5 days a week for 12 weeks. The MovAlyzeR® keeps track (records) all the participants' practice. MovAlyzeR is HIPPA compliant. We use the MovAlyzeR as a training device for handwriting, not for data collection. Since MovAlyzeR provides instant feedback to the user on their handwriting movement, it is a fun way for the children to practice handwriting.
Masking Description: Participant will practice 5 days p/week, 15-20 minutes p.day for 12 weeks. They will receive only feedback from the software program as they practice handwriting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Participants are diagnosed with tic disorder and/or Tourette syndrome. They will undergo treatment to improve overall handwriting skills.
  Interventions: Other: Handwriting intervention

INTERVENTIONS:
Other: Handwriting intervention — children will practice handwriting 5 days p/week, 15-20 minutes p/day for 12 weeks using the movalyzer software program.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a computerized handwriting training protocol (MovAlyzeR), through daily practice of handwriting on an electronic device to improve handwriting skills in children with tic disorders (TD).

DETAILED DESCRIPTION:
Handwriting is a functional skill underlying almost all academic performance of school-aged children, and handwriting impairment is highlighted by the World Health Organization as a barrier to school participation. The available evidence mentioned in the literature suggests handwriting skills are academically crucial, and handwriting deficits may lead to challenges in performing various academic activities both in and outside the classroom.

Given that children with TD are more likely to have handwriting deficits as suggested in a recent study, they are also more likely to have challenges in their academic performance and success as evidenced in the literature.

In the context of education, strong evidence indicated that handwriting has more cognitive and neurological benefits than using a keyboard when taking notes in the classroom. Therefore, reducing tics and improving handwriting skills rather than an adaptation approach using a word processor or computer may be the goal of intervention.

Results of the investigator's previous study showed that children with Tourette Syndrome (TS) or tic disorders (TD) demonstrated handwriting deficits when compared to the general children population, and were consistent with a recent study conducted in France showing that children with TS exhibited handwriting problems. In addition to illegibility issues in handwriting as indicated by the low score on the Test of handwriting skills (THS-R), children with TS or TD also demonstrated writing deficits in the areas of speed of writing and correct letter case formation.

Since handwriting deficit is an area of concern among children with TS or TD, one way to improve these children's handwriting skills is through handwriting practice. NeuroScript, LLC., has developed a software program (MovAlyzeR) that allows children to practice handwriting on an electronic device (such as tablet, laptop, etc). Given that the practice is completed on an electronic device with immediate feedback, this handwriting program may serve as a strong incentive to motivate children practicing handwriting. In order to provide evidence for the educators and therapists on the effectiveness of this software program, it is important to evaluate its effectiveness on improving handwriting skills among children with TS or TD.

ELIGIBILITY:
Inclusion Criteria:

* Tourette syndrome
* Diagnosed tic disorder

Exclusion Criteria:

* Diagnosed anxiety disorder
* Diagnosed learning disability
* Diagnosed dysgraphia

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Scores of handwriting competence for legibility | Pre treatment, baseline
  Scores are recorded by standard scores. Children scoring greater than 1 standard deviation below the mean of 100 will receive intervention.
Scores of handwriting competence for legibility | Post treatment, after week 12
  Scores are recorded by standard scores with a mean of 100.
Scores of handwriting competence for speed | Pre treatment, baseline
  Scores are recorded by standard scores. Children scoring greater than 1 standard deviation below the mean of100 will receive intervention.
Scores of handwriting competence for speed | Post treatment, after week 12
  Scores are recorded by standard scores with a mean of 100
Percentage of handwriting competence for reversal of letters | Pre treatment, baseline
  Reversal of letters are scored as an ancillary score using three categorizations: test further (i.e., below 16th percentile or more one standard deviation (SD) below the normative mean or z-score < -1), watch (i.e., between 16th percentile and 50th percentile), and no concern (i.e., 50th percentile and above). Children scoring below 16% or 1 standard deviation below will receive intervention.
Percentage of handwriting competence for reversal of letters | Post treatment, after week 12
  Reversal of letters are scored as an ancillary score using three categorizations: test further (i.e., below 16th percentile or more one standard deviation (SD) below the normative mean or z-score < -1), watch (i.e., between 16th percentile and 50th percentile), and no concern (i.e., 50th percentile and above).
Percentage of handwriting competence for letters touching one another | Pre treatment, baseline
  Letters touching each other are scored as an ancillary score using three categorizations: test further (i.e., below 16th percentile or more one standard deviation (SD) below the normative mean or z-score < -1), watch (i.e., between 16th percentile and 50th percentile), and no concern (i.e., 50th percentile and above). Children scoring below 16% or 1 standard deviation below will receive intervention.
Percentage of handwriting competence for letters touching one another | Post treatment, after week 12
  Letters touching each other are scored as an ancillary score using three categorizations: test further (i.e., below 16th percentile or more one standard deviation (SD) below the normative mean or z-score < -1), watch (i.e., between 16th percentile and 50th percentile), and no concern (i.e., 50th percentile and above).
Percentage of handwriting competence for case errors | Pre treatment, baseline
  Case errors are scored as an ancillary score using three categorizations: test further (i.e., below 16th percentile or more one standard deviation (SD) below the normative mean or z-score < -1), watch (i.e., between 16th percentile and 50th percentile), and no concern (i.e., 50th percentile and above). Children scoring below 16% or 1 standard deviation below will receive intervention.
Percentage of handwriting competence for case errors | Post treatment, after week 12
  Case errors are scored as an ancillary score using three categorizations: test further (i.e., below 16th percentile or more one standard deviation (SD) below the normative mean or z-score < -1), watch (i.e., between 16th percentile and 50th percentile), and no concern (i.e., 50th percentile and above).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Rowe, Dr OT, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined